CLINICAL TRIAL: NCT01428700
Title: Development of Gene Expression Signatures for the Diagnosis of Liver Allograft Rejection and Recurrent Hepatitis C Disease (CTOT-07)
Brief Title: Gene Expression in Liver Allograft Rejection and Recurrent Hepatitis C
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOT-07
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Liver tissue, whole blood, and serum specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-Immune/Non-Viral (NINV): Patients enrolled in ITN030ST transplanted for liver failure resulting from non-viral, non-immune causes
- Hepatitis C Virus (HCV) positive: Patients enrolled in ITN030ST transplanted for liver failure resulting from HCV genotype 1 infection

SUMMARY:
Acute cellular rejection is relatively common after liver transplantation, typically does not affect graft survival, and is not associated with the development of chronic rejection. Acute cellular rejection is diagnosed when liver enzymes and/or liver function tests are elevated when compared to baseline. The only means of differentiating acute rejection from other liver pathologies is with a liver biopsy. However, even with this invasive diagnostic procedure, it may be difficult to distinguish acute rejection from another disease process, such as injury caused by the hepatitis C virus (HCV) from the native liver. This study will evaluate whether certain patterns of biomarkers in the peripheral blood and/or liver tissue of a liver transplant recipient can be used to determine if the transplanted liver is being rejected by the recipient or sustaining HCV injury. Diagnostic biomarkers that are specific for acute rejection and informative of the severity of HCV recurrence could allow for modulation of immunosuppression therapy and treat the clinical condition without the need for invasive liver biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Specimens derived from subjects enrolled in the ITN030ST study.
* Availability of adequate biopsy specimens with corresponding blood and/or serum collected within a 10 day window of a for-cause or protocol biopsy.

Exclusion Criteria:

* Withdrawal of consent for the ITN030ST study.
* Absence of consent in the ITN030ST study for the collection and storage of samples of blood and tissue for future research studies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled in ITN030ST (NCT00135694)
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Expression levels of mRNA and miRNA in peripheral blood cells, serum, and tissue at the time of for cause and protocol biopsies, and the diagnostic effectiveness of identified patterns | +/- 10 day window from time of clinically indicated biopsy
  This assay study will analyze expression levels of mRNA and miRNA from NINV and HCV liver biopsy, whole blood, and/or serum samples from the ITN030ST study obtained within a +/- 10-day window of the biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Shaked, MD, PhD, Principal Investigator — University of Pennsylvania; Manikkam Suthanthiran, MD, Study Chair — Cornell University

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/
- See also: Clinical Trials in Organ Transplantation (CTOT) — https://www.ctotstudies.org/